CLINICAL TRIAL: NCT01128608
Title: The Effect of High PCO2 Solution on Esophageal Acid Sensation in Healthy Patients Versus Those With Non-Erosive Reflux Disease.
Brief Title: The Effect of High PCO2 Solution on Esophageal Acid Sensation
Acronym: PC02
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southern Arizona VA Health Care System (U.S. Federal Agency)
Responsible Party: Ronnie Fass, M.D., Southern Arizona VA Health Care System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: The Effect of PCO2 Solution
Record Dates: First submitted 2010-05-21; First posted 2010-05-24 (Estimated); Last update posted 2010-07-21 (Estimated); Status verified 2010-04

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: GERD; Heartburn; Acid Reflux
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group - Healthy Subjects (Active Comparator): Healthy volunteers with normal EGD.
  Interventions: Procedure: PCO2 Acid Perfusion and 0.1N HCI Perfusion
- NERD Group (Active Comparator): Subjects with NERD. Heartburn symp x2 wk for 3 months. Normal EGD and abnormal 24 hour pH.
  Interventions: Procedure: 24-Hr Esohpageal pH Monitoring

INTERVENTIONS:
Procedure: 24-Hr Esohpageal pH Monitoring — There will be a 24-hr pH monitoring procedure and two 10-minute infusions each one week apart consisting of high PCO2 solution and 0.1 N HCI solution.
  Arms: NERD Group
Procedure: PCO2 Acid Perfusion and 0.1N HCI Perfusion — A small tube will be inserted through the nostril and into the esophagus. A mild CO2 solution or a mild saline solution will be administered for aprox. 10 minutes during which you will be asked questions regarding any symptoms you may experience.
  Arms: Control Group - Healthy Subjects

SUMMARY:
To determine the effect of intraesophageal high PCO2 solution as compared to acidic and saline solutions on subjects' heartburn sensation using stiumlus-response functions.

DETAILED DESCRIPTION:
Presently, the exact mechanism of GERD and the role of CO2 in pathogenesis of heartburn symptoms is unclear. CO2 conversion to protons may play a key role in the mechanism for heartburn sensation. This is a prospective, randomized study that will help further explore the mechanism for heartburn sensation in GERD patients and can be a prelude for further studies examining the role of new class antireflux agents such as carbonic anhydrase inhibitors in the treatment of patients with heartburn.

ELIGIBILITY:
Inclusion Criteria:

10 Healthy Controls

* Normal EGD, Normal 24-hr pH
* 18-80 Years of age
* Able to read, understand and complete study questionnaires and diary
* Able to understand study procedures and sign informed consent
* Albe to comply with all study requirements

  10 NERD (Non-Erosive Reflux Disease)
* 18-80 Years of age
* Willing to stop PPI/H2 Blocker prior to EGD
* Have heartburn symptoms 2+ times per week for at least 3 months.

Exclusion Criteria:

* Esophageal erosions, Barretts, or peptic stricture on EGD
* Previous esophageal, gastric or duodenal surgery
* underlying co-morbidities
* Diabetes mellitus (requires insulin), scleroderms, or neuromuscular disorder
* Upper airway symptoms
* Tricyclic antidepressants, antispasmodics, selective serotonin receptor inhibitors, thiazides, bile acid-binding agents or prokinetics
* Patients who cannot or are unwilling to sign ICF

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-10 (Estimated); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
The Mechanism of GERD | NA There is no exact timeframe.
  Presently the exact mechanism of GERD and the role of CO2 in pathogenesis of heartburn sysmptoms is unclear. We aim to compare the effect of intraesophageal high PCO2 solution with saline solution on heartburn sensation.

CONTACTS AND LOCATIONS:
Overall Officials: Ronnie Fass, MD, Principal Investigator — Southern Arizona Veterans Health Care System
Locations (2):
- United States (2):
  - Southern Arizona VA Health Care System, Tucson, Arizona
  - Southern Arizona Veterans Health Care System, Tucson, Arizona